CLINICAL TRIAL: NCT06486025
Title: ALTERNATE DOSING PROTOCOL FOR MAGNESIUM SULFATE IN OVERWEIGHT AND OBESE WOMEN WITH PREECLAMPISA: A RANDOMIZED CONTROLLED TRIAL
Brief Title: Protocols for Magnesium Sulfate Maintenance Dose in Overweight and Obese Women Diagnosed With Preeclampsia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Magnesium and Preeclampsia
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Severe Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium Sulphate 1g/hr (Active Comparator): Women in this group will receive a routine loading infusion of 5 g of MgSO4 over 20 minutes, followed by a maintenance dose rate of 1 g/h.
  Interventions: Drug: maintenance magnesium sulphate1g/h
- Magnesium Sulphate 2g/hr (Active Comparator): Women in this group will receive a routine loading infusion of 5 g of MgSO4 over 20 minutes, followed by a maintenance dose rate of 2 g/h.
  Interventions: Drug: maintenance magnesium sulphate2g/h

INTERVENTIONS:
Drug: maintenance magnesium sulphate1g/h — Women will receive a routine loading infusion of 5 g of MgSO4 over 20 minutes, followed by a maintenance dose rate of 1 g/h.
  Arms: Magnesium Sulphate 1g/hr
Drug: maintenance magnesium sulphate2g/h — Women will receive a routine loading infusion of 5 g of MgSO4 over 20 minutes, followed by a maintenance dose rate of 2 g/h.
  Arms: Magnesium Sulphate 2g/hr

SUMMARY:
There is still no evidence of the appropriate dose to be used. Serum magnesium sulfate concentration is not measured regularly, thus we may be using sub-therapeutic level or reaching a toxic level.Overweight and obese women have different pharmacokinetics and different drug distribution, therefore, they may need higher doses of magnesium sulfate to reach therapeutic level.

DETAILED DESCRIPTION:
Magnesium sulfate is used in pre-eclampsia to prevent seizures, it is administered in the form of a loading dose and maintenance dose. Maintenance dose of magnesium sulfate in pre-eclampsia varies in literature (1-3gms/hour). There is still no evidence of the appropriate dose to be used. Serum magnesium sulfate concentration is not measured regularly, thus we may be using sub-therapeutic level or reaching a toxic level.Overweight and obese women have different pharmacokinetics and different drug distribution, therefore, they may need higher doses of magnesium sulfate to reach therapeutic level. This study will evaluate whether overweight and obese women need higher maintenance doses to reach therapeutic level of magnesium sulfate in serum.Preeclampsia is a serious pregnancy complication characterized by hypertension, proteinuria and signs of damage to another organ system, often the kidneys, occurring after 20 weeks of gestation

ELIGIBILITY:
Inclusion Criteria:

Women diagnosed with SPET as per criteria of NICE, 2023 guidance

* Age 20-40 years
* BMI >25kg/m2
* Gestational age > 28 weeks

Exclusion Criteria:

* Intrauterine Fetal Death (IUFD)
* Hemolysis - Elevated liver enzymes - Low platelets syndrome (HELLP)
* Contraindication to Magnesium Sulfate such as myasthenia gravis, severe renal failure, cardiac ischemia, and heart block
* Serum creatinine levels greater than 1.1 mg/dL.
* Women refusing to participate in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
serum magnesium level | 24 hours
  Maternal Serum Magnesium Level after 24 hours of magnesium sulphate infusion